CLINICAL TRIAL: NCT04724772
Title: Comparison of Clinical Outcomes Following Upper Lid Blepharoplasty With and Without Tranexamic Acid as an Additive to Traditional Local Anesthetic.
Brief Title: Use of Tranexamic Acid in Blepharoplasties
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped study due to pharmacy issues before treating patients
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Douglas Sidle, Investigator, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STU00211373
Record Dates: First submitted 2021-01-05; First posted 2021-01-26 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Pain, Postoperative; Bruising
MeSH Terms: conditions — Pain, Postoperative; Contusions | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Each patient is blinded to which eye receives TXA. All patients have both eyes injected with LA, and one eye injected with TXA.
Masking Description: The patient does not know which side receives the TXA in addition to the LA. They then personally assess pain and bruising. The provider is blinded to which syringe has both TXA and LA, and which only has LA.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blepharoplasty patient (Experimental): Patient receives LA in one eye and LA with TXA in the other eye. They are blinded. They compare eyes without knowing which one received the TXA.
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: Tranexamic acid injection — Injection of tranexamic acid preoperatively

SUMMARY:
The goal of this investigation is to assess whether or not there is a significant difference in the presence and/or degree of post-operative ecchymosis, pain, and edema between groups of patients undergoing upper lid blepharoplasty with traditional local anesthetic (LA) and those who receive tranexamic acid (TXA) in addition to traditional LA.

DETAILED DESCRIPTION:
Blood clot formation involves a cascade of reactions that results in the production of thrombin, which converts fibrinogen into fibrin. In turn, fibrin aggregates and forms a clot. Hemostasis depends on a balance between this clotting cascade and the processes that break down clots, particularly the conversion of plasminogen to plasmin and plasmin's subsequent degradation of fibrin polymers. Tranexamic acid (TXA) is an agent, first patented in 1957, that competitively inhibits plasmin generation and activity.

As a result, TXA promotes clotting and, therein, hemostasis, making it useful for controlling surgical bleeding. (See figure below.) Indeed, a 2012 meta-analysis demonstrated that administering TXA intra- or perioperatively reduces the probability of receiving a blood transfusion by one-third.

Additionally, large trials have shown that TXA does not increase the risk of thromboembolic events in patients. One study noted that there was a slightly increased incidence of seizures in patients who received TXA, though this was limited to patients who underwent open-heart surgery, which is, itself, an independent risk factor for seizures. Another study halved the dose of TXA administered to its participants, but this did not reduce seizure risk amongst the participants. Thus, the data on this adverse effect remains inconclusive, and surgeons continue using TXA for its hemostatic effects, especially in cardiac and orthopedic surgeries. Given that facial plastic surgery does not incur the same sort of blood loss as cardiac or orthopedic surgery, efforts to describe TXA use in this field have focused on its established anti-inflammatory properties in addition to hemostasis. There are reports of TXA use in rhinoplasties, face lifts, and blepharoplasties; however, such reports are scarce, with randomized, double-blinded, controlled clinical trials even more so. Only one study has examined TXA use in blepharoplasties. In that study, 34 patients were randomized to receive an injection of lidocaine mixed with either TXA or saline. The authors did not find any significant difference in post-operative parameters including size of periocular ecchymoses and patient-reported pain level. Since the only randomized controlled trial investigating TXA use in blepharoplasty involved 34 participants, the investigators aim to add to the body of knowledge on this matter.

Furthermore, the investigator's study will be structured differently from that of Sagiv et al. Firstly, the patients will serve as their own controls, since we will inject one eyelid with a solution containing TXA and another with a placebo solution. This will help reduce bias between study groups that may have existed in Sagiv et al's trial. Secondly, the investigators will follow the patients for 3 months after the procedure, which is eleven weeks longer than the duration of follow-up amongst participants in Sagiv et al's trial. This will give the investigators an even better sense of TXA's impact on patients' post-operative courses. In summary, the investigators wish to characterize TXA's hemostatic and anti-inflammatory effects in patients who undergo blepharoplasty. Since there is currently only one publication that accomplishes this, the investigators' objective is to expand knowledge in this area so that surgeons performing facial plastic procedures can optimize patients' recovery and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* any adult patient who is undergoing upper lid blepharoplasty with author Douglas Sidle, MD and who is older than 18 years of age, fluent in English, not on any anticoagulant or antiplatelet medication (e.g. aspirin, clopidogrel, etc.), not diagnosed with a coagulation disorder, not pregnant, not undergoing a simultaneous procedure, and not a Feinberg School of Medicine (FSM) student or Northwestern Memorial (NM) employee.

Exclusion Criteria:

* less than 18 years of age, not fluent in English, taking anticoagulant or antiplatelet, has coagulation disorder, pregnant, simultaneous procedure, FSM or NM student/employee

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2023-07-20 (Estimated); Study Completion 2023-09-20 (Estimated)

PRIMARY OUTCOMES:
change in bruising | Surveys will be completed by patients at 1 week, 1 month, 3 months post-operatively
  patients are given a survey to rate bruising on each side, change will be assessed from different time periods
change in bruising a survey to rate pain | Surveys will be completed by patients at 1 week, 1 month, 3 months post-operatively
  patients are given a survey to rate pain on each side, change will be assessed from different time periods

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No